CLINICAL TRIAL: NCT01295567
Title: Can Dipyridamole Induce Protection Against Ischemia and Reperfusion Injury in Patients Undergoing Elective CABG?
Brief Title: Can Dipyridamole Induce Protection Against Ischemia and Reperfusion Injury in Patients Undergoing Elective Coronary Artery Bypass Grafting (CABG)?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, G. Rongen, professor, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dipy-cabg; 2009-014299-22 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-14 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Disease; Ischemic Heart Disease
Keywords: ischemia reperfusion injury; CABG; dipyridamole; HS-troponin-I
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia; Reperfusion Injury | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- dipyridamole (Experimental)
  Interventions: Drug: Dipyridamole

INTERVENTIONS:
Drug: Dipyridamole — prior to CABG surgery 3 day treatment with dipyridamole 200mg SR twice daily
  Other Names: persantin
  Arms: dipyridamole
Drug: placebo — prior to CABG surgery 3 day treatment with placebo capsules twice daily
  Arms: placebo

SUMMARY:
Rationale:

Due to western lifestyle human coronary arteries are prone to develop atherosclerotic plaques. Hence the heart is an important target organ for atherothrombotic complications: myocardial ischemia, arrhythmias, myocardial infarction and heart failure. To alleviate symptoms and decrease mortality in these patients, myocardial revascularisation is recommended. Coronary artery bypass grafting (CABG) is indicated in patients with severe atherosclerotic disease of all three coronary arteries or the left main stem coronary artery. Cardiac ischemia and reperfusion injury during CABG is inevitable and jointly accountable for complications that occur after CABG (e.g. death, myocardial infarction, arrhythmias, stroke, or renal complications). Dipyridamole has been shown to reduce ischemia reperfusion injury in healthy volunteers using an intermediate endpoint and may prevent cardiovascular death or event in secondary prevention after cerebrovascular disease. The investigators hypothesise that oral pre-treatment with dipyridamole can increase cardiac tissue tolerance against ischemia and reperfusion injury due to CABG. The investigators expect lower troponin-I release in patients who were pretreated with dipyridamole.

Objective: To study the effect of oral pretreatment with dipyridamole on high sensitivity (HS)-troponin-I release after CABG. Secondary objectives are whether oral pretreatment with dipyridamole reduces postoperative CABG arrhythmias, prolonged inotropic support, and duration of Intensive Care-stay. Further secondary endpoints are the effects of dipyridamole pretreatment on renal injury and post-ischemic recovery of contractile function (measured ex-vivo).

Hypothesis:

The investigators hypothesize that oral pre-treatment with dipyridamole can increase cardiac tissue tolerance against ischemia and reperfusion injury. The investigators expect lower HS-troponin-I release in patients who were pretreated with dipyridamole. Additionally the investigators expect the incidence of arrhythmias, need for prolonged inotropic support (longer than 24 hours postoperative) to be decreased in pretreated patients.

ELIGIBILITY:
Inclusion Criteria:

* Acceptation for CABG in RUNMC
* Informed consent

Exclusion Criteria:

* Recent myocardial infarction (STEMI or non-STEMI), during two weeks prior to inclusion
* Asthma
* Use of insulin
* Use of sulfonylurea derivates (e.g. glibenclamide, tolbutamide, gliclazide, glimepiride)
* Use of metformin
* Use of oral corticosteroids
* Use of dipyridamole
* Use of clopidogrel within 8 days prior to scheduled CABG surgery
* Chronic use of Non Steroid Anti-Inflammatory Drugs (NSAIDs)
* Off-pump surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HS-troponin-I | within 72 hours after CABG.
  high sensitivity cardiac troponin-I

SECONDARY OUTCOMES:
duration of inotropic support | within three days after CABG
duration of IC stay | within three days after CABG
drain production | 24 hours after surgery and total drain production within three days after surgery
  thoracic drain production after CABG
post-ischemic recovery of contractile function | until 4 hours after harvesting
  The right atrial appendage is harvested during cardiac surgery before the introduction of the extracorporal circulation. Two atrial trabeculae are dissected, suspended in an organ bath, and linked to a force transducer. after equilibration and baseline measurement, simulated ischemia and reperfusion influences contractile force recovery
Renal damage | Within three days after CABG
  biomarkers for renal failure will be detemined in blood and urine before and after CABG

CONTACTS AND LOCATIONS:
Locations (1):
- RUNMC, Nijmegen, Netherlands

REFERENCES:
- [Derived] El Messaoudi S, Wouters CW, van Swieten HA, Pickkers P, Noyez L, Kievit PC, Abbink EJ, Rasing-Hoogveld A, Bouw TP, Peters JG, Coenen MJ, Donders AR, Riksen NP, Rongen GA. Effect of dipyridamole on myocardial reperfusion injury: A double-blind randomized controlled trial in patients undergoing elective coronary artery bypass surgery. Clin Pharmacol Ther. 2016 Apr;99(4):381-9. doi: 10.1002/cpt.106. Epub 2015 Oct 22. PMID 25773594